CLINICAL TRIAL: NCT05439954
Title: Application of MRI Radiomics to Improve Diagnosis and Pharmacologica Prognosis of Autism Spectrum Disorder
Brief Title: Radiomics of Autism Spectrum Disorder
Status: Active, not recruiting | Type: Observational
Sponsor: Qingling Chen (Other)
Responsible Party: Sponsor-Investigator, Qingling Chen, Doctor, Fifth Affiliated Hospital, Sun Yat-Sen University
Organization: Fifth Affiliated Hospital, Sun Yat-Sen University (Other)
Other Study IDs: QL Chen
Record Dates: First submitted 2022-06-27; First posted 2022-06-30 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Autism Spectrum Disorder
Keywords: MRI; radiomics
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case group: （a）patients fulfilling the Diagnostic Criteria of the Diagnostic and Statistical Manual of Mental Disorders 5th Edition（DSM-V); (b)age:14 and under 14 years old; (c)first clinic visit, never-treated; (d)without injury to head and other diseases of the nervous system.
- Control Group: （a）healthy subject of same ages;(b)without injury to head and diseases of the nervous system; (c)without family history of mental disorders; (d)without other somatic illness.

SUMMARY:
Autism Spectrum Disorder (ASD) refers to a group of neurodevelopmental disorders including autism.Despite ongoing studies, the pathogenesis of ASD still remains unclear.The global prevalence of ASD was estimated at 1% in 2015.The diagnostic criteria for ASD are specified in the DSM ( American Psychiatric Association, 2013 ) and serve as guideline for clinicians at the present. However, its early diagnosis value is limited due to a high subjectivities and its low diagnostic sensitivity and specificity.Early detection and early pharmacological and behavioral interventions are critical in improving the symptoms and preventing the disease progression. There are no medications that directly treat the core symptoms present in individuals with ASD, and the effectiveness of interventions remains limited. Therefore, accurate assessment of pharmacological efficacy is necessary for the reatment, and prognostication of individuals with ASD. Magnetic resonance imaging (MRI) is a commonly used imaging tool for clinical disease diagnosis, especially for neurological disorders. Besides, Structural Magnetic Resonance imaging reflects neuropathological and microstructural developmental changes during growth. Radiomics based on the high-dimensional quantitation of medical images, allowing extraction of more detailed characteristics than is possible with conventional visual interpretation. This study aims: (1)To explore an objective diagnostic method through radiomics in children with ASD (2)to provide prognostic estimates of the outcome, based on estimates of an individual patient's prognosis and the efficacy of different drug therapies.

ELIGIBILITY:
Inclusion Criteria:（a）healthy subject of same ages;(b)without injury to head and diseases of the nervous system; (c)without family history of mental disorders; (d)without other somatic illness.

Exclusion Criteria:

-

Ages: 1 Year to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: （a）patients fulfilling the Diagnostic Criteria of the Diagnostic and Statistical Manual of Mental Disorders 5th Edition（DSM-V); (b)age:14 and under 14 years old; (c)first clinic visit, never-treated; (d)without injury to head and other diseases of the nervous system.
Sampling Method: Non-Probability Sample
Enrollment: 230 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
diagnosis of autism spectrum disorder | 01/12/2022
  differential diagnosis of case group and control group

CONTACTS AND LOCATIONS:
Locations (1):
- The Fifth Affiliated Hospital at Sun Yat-sen University, Zhuhai, Guangdong, China

IPD SHARING:
Plan to Share IPD: No